CLINICAL TRIAL: NCT03961282
Title: CODY (Co-design for You): An Immersive Technology Tool for Experiencing and Assessing Home Alterations for Veterans With Movement Disabilities and Disorders
Brief Title: CODY (Co-design for You): An Immersive Technology Tool for Experiencing and Assessing Home Alterations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201802634
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Parkinson Disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: There are 3 types of door alterations in a simulated residential setting being tested: Standard (conforms to conventional residential building practices); Enhanced (conforms to Americans with Disabilities Act or ADA residential building practices or recommendations); and Co-design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson Disease Group (Experimental): Each participant is randomized into 3 types of door alterations: Standard (conforms to conventional residential building practices); Enhanced (conforms to Americans with Disabilities Act or ADA residential building practices or recommendations); and Co-design. Then each participant performs Test #1: Doorway Width and Test #2: Door Frame Color.
  Interventions: Other: Doorway Width Test; Other: Door Frame Color Test
- Healthy Participant Group (Experimental): Each participant is randomized into 3 types of door alterations: Standard (conforms to conventional residential building practices); Enhanced (conforms to Americans with Disabilities Act or ADA residential building practices or recommendations); and Co-design. Then each participant performs Test #1: Doorway Width and Test #2: Door Frame Color.
  Interventions: Other: Doorway Width Test; Other: Door Frame Color Test

INTERVENTIONS:
Other: Doorway Width Test — The first test consists of Doorway Width. Standard level is a doorway width of 30 inches; Enhanced is doorway width of 36 inches; Co-design allows the participant to adjust the width anywhere from 26 to 48 inches.
  Other Names: Test #1
Other: Door Frame Color Test — The second test consists of Door Frame Color. Standard level is same color (hue) as light-color wall; Enhanced level is same hue but of higher color intensity for contrast; Co-design allows the participant to adjust the color intensity range from lowest (same as wall) to highest intensity (stronger contrast than in Enhanced).
  Other Names: Test #2

SUMMARY:
CODY (co-design for you) is a Virtual Reality (VR) tool and Application Programming Interface (API) which uses an immersive, interactive environment for using, experiencing and co-designing home alterations. The aim of this research is to assess the efficacy of using CODY to aid and enhance the ability of adults with Parkinson's disease (PD) to experience and choose appropriate home modifications.

DETAILED DESCRIPTION:
Accessible housing is a widespread need in this country. This is particularly true among those persons with mobility impairments and movement disorders. While design and construction guidebooks exist for modifying homes for people with disabilities, there are also many documented instances where a standard, "by-the-book" alteration or assistive technology did not support the need or condition of the particular individual it was intended for. Just as occupational therapists recognize that a critical component of successful rehabilitation assistance is a person-centered plan that facilitates individualized solutions, likewise diverse design (or home alterations/modification, referred here as HM) approaches which approximate a person-centered plan also provide a more effective fit for persons with disabilities. A "one-size-fits-all" approach is not comprehensive for the diverse disability community.

This research entails the design and development of CODY (co-design for you), a Virtual Reality (VR) tool and Application Programming Interface (API), which uses an immersive, interactive environment for using, experiencing and co-designing home alterations. The 'co-design' nature of CODY denotes that persons with movement disorders, such as Parkinson's disease can: virtually interact with and experience a home alteration/modification (HM) in a virtual, simulated environment; have multiple variations of a HM that the user can choose from; and is able to assess and manipulate the HM for appropriateness to one's need and circumstances before actually installing devices or making modifications to one's own home. As such, CODY is a new assistive technology that aids and enhances the ability of individuals with disabilities to live in adapted homes that supports their needs.

This study focuses on movement disorders faced by persons with Parkinson's disease (PD) to demonstrate how effective CODY may be for those with major movement challenges, characterized by tremor, bradykinesia, postural instability, and freezing of gait (FoG). Collectively, these symptoms increase fall risk, fear of falling and impact the quality of life when compared to other age-matched non-PD adults. While clinical observations suggest that attributes of the physical interior environment may make daily activities easier or harder for persons with PD, few studies have actually examined the impact of specific changes in interior design on an individual's performance. One research study revealed that FoG, one of the major contributors to falls, was induced by doorways. Another study similarly revealed a significant increase in doorway-provoked FoG indicators by decreasing doorway width.

The aims of this research are: (1) To develop the Virtual Reality-based CODY tool and corresponding API; and (2) To assess the efficacy of using CODY to aid and enhance the ability of persons with PD to experience and choose appropriate home modifications. The underlying purpose of CODY is to provide opportunities for the growing population of persons with movement disabilities and disorders to actively engage in decisions affecting their living environment. Although VR games have been used for rehabilitation and therapy purposes, no research studies exist that demonstrate the use or effectiveness of integrated VT simulations in allowing persons with disabilities to interactively design residential alterations. The study team's expectation is that CODY will not only be successful in this short-term pilot study, but will lead to further refinement, development and, potentially, a commercial product. The investigators envision CODY's integrated, immersive, and interactive simulation will be used by neurologists, rehabilitation specialists, and occupational therapists for working with consumers to assess and determine optimal home modifications for those with ambulatory and other movement impairments.

ELIGIBILITY:
Inclusion Criteria: Parkinson's Disease participants

* Patients with a mild-to-moderate diagnosis of PD, evaluated using the Unified Parkinson's Disease Rating Scale (UPDRS) and the Modified Hoehn and Yahr stages I-III, by a fellowship trained neurologist, arriving at the diagnosis by applying strict UK Brain Bank criteria
* Disease duration is less than 5 years
* With phone area code of 352; 904
* Currently on their medications Inclusion Criteria: Healthy participants
* Individuals who indicated they would like to be contacted for future research opportunities.
* Age-matched (+ or - 5 years) healthy participants without PD
* No history of neurological or orthopedic problems that could impair walking function or upper extremity mobility

Exclusion Criteria:

* Individuals with atypical features of PD, peripheral neuropathy, vestibular dysfunction, and medications affecting balance or alertness/ attention
* Individuals with the presence of active unstable medical, diabetes, or any orthopedic conditions
* Individuals who have previously undergone any brain surgeries
* Individuals who take any anti-psychotic medications
* Individuals with dementia as reflected by performance on the Mini-Mental State Examination (MMSE) (score < 24)
* Individuals with elevated scores on the Beck Depression Inventory-II (I.E., ≥20), the recommended cut-off for depressive symptoms in PD by the task force for the Movement Disorders Society or history of severe pre-existing psychiatric difficulties (i.e., schizophrenia)

Ages: 40 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Gait time | Day 1 (3 seconds)
  Participant will be instructed to walk on a 8' 6" long gait mat and pass through the doorway seen on the headset display. The middle portion of the gait mat with a length of 4' 3" is pressure sensitive and transmits gait time data to the software installed in the encrypted desktop. Gait time is the time between the first heel strike and the last toe off on the mat during the walk is measured as gait time.
Step time | Day 1 (0.8 second)
  Participant will be instructed to walk on a 8' 6" long gait mat and pass through the doorway seen on the headset display. The middle portion of the gait mat with a length of 4' 3" is pressure sensitive and transmits step time data to the software installed in the encrypted desktop. Step time is the time to complete one full gait cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Srinivasan, PhD, Principal Investigator — University of Florida; Shabboo Valipoor, PhD, Principal Investigator — University of Florida
Locations (1):
- Shimberg Center for Housing Studies, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No